CLINICAL TRIAL: NCT02114619
Title: The Effect of Different Calculated Doses of I-131 in Treatment of Patients With Grave's Disease
Brief Title: Comparative Study of Different I-131 Doses in Graves' Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, S.R.ZAKAVI, Head of Nuclear Medicine Research Center, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 920800
Record Dates: First submitted 2014-04-12; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Graves' Disease
Keywords: radioiodine therapy; Graves' disease; Hyperthyroidism; calculated dose
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — Iodine-131

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose of I-131 (Active Comparator): Patients with Graves' disease who will be treated with I-131, using 100 microcurie per gram (uCi/gr) of thyroid weight
  Interventions: Drug: Low dose of I-131
- Intermediate dose (Active Comparator): Patients with Graves' disease who will be treated with 150 microcurie (uCi) of I-131 per gram of thyroid weight.
  Interventions: Drug: Intermediate dose
- High dose (Active Comparator): Patients with Graves' disease who will be treated with I-131 using 200 uCi/gr of thyroid weight.
  Interventions: Drug: High dose

INTERVENTIONS:
Drug: Low dose of I-131 — We wil administer 100 micro currie of iodine per thyroid gram
  Arms: Low dose of I-131
Drug: Intermediate dose — We will administer 150 micro currie of iodine per thyroid gram
  Arms: Intermediate dose
Drug: High dose — We will administer 200 micro currie of iodine per thyroid gram
  Arms: High dose

SUMMARY:
Radioactive iodine (RAI) administration is an effective and completely established treatment modality in hyperthyroidism including Graves' disease. Despite the long experience with radioiodine for hyperthyroidism, controversy remains regarding the optimal dose of iodine that is required to achieve long-term euthyroidism. The fixed activity administration method does not optimize the therapy, giving often too high or too low radiation to the gland, but the optimal dose per gram of thyroid mass in calculated activity administration method is also under much debates. This prospective study has been designed in order to compare the effect of different calculated doses of radioiodine on Graves' disease treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 hyperthyroid patients (Graves'disease)

Exclusion Criteria:

* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
change of thyroid related hormones blood level from baseline at 1,3,6 and 12 month | 1,3,6,12 month
  thyroid-stimulating hormone (TSH), T4, T3

SECONDARY OUTCOMES:
Rate of hypothyroidism status at 1, 3,6 and 12 month post RAI therapy | 1,3,6,12 month
  Hypothyroidism index

OTHER OUTCOMES:
Change of thyroid volume | 1,3,6 and 12 months
  Change of thyroid volume 1,3,6 and 12 months after therapy using ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Narjess Ayati, MD, FEBNM, Study Director — Nuclear Medicine Research Center
Locations (1):
- Nuclear Medicine Research Center, Ghaem Hospital, Mashhad, Khorasan-Razavi, Iran